CLINICAL TRIAL: NCT05073003
Title: A Staged Phase I/II Observer-blind, Randomised, Controlled, Multi-country Study to Evaluate the Safety, Reactogenicity, and Immune Responses to the GVGH altSonflex1-2-3 Vaccine Against S. Sonnei and S. Flexneri, Serotypes 1b, 2a, and 3a, in Adults in Europe (Stage 1) Followed by Age De-escalation From Adults to Children and Infants, and Dose-finding in Infants in Africa (Stage 2)
Brief Title: A Study on the Safety and Immune Responses to the GVGH altSonflex1-2-3 Vaccine Against Shigellosis in Adults, Children, and Infants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 212149; 2021-000891-12 (EudraCT Number)
Record Dates: First submitted 2021-09-29; First posted 2021-10-11 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Diarrhoea
Keywords: Shigella infection; Shigellosis; Diarrhoea; S. sonnei; S. flexneri; Low and middle income countries
MeSH Terms: conditions — Diarrhea; Dysentery, Bacillary | interventions — Shigella Vaccines; Meningococcal Vaccines; Boostrix; Tetanus Toxoid; Hepatitis B Vaccines; diphtheria-tetanus-acellular pertussis-inactivated poliovirus-Haemophilus influenzae b conjugate-hepatitis B vaccine; Vi polysaccharide vaccine, typhoid; Rubella Vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Observer blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (20):
- ST1_Adults_Placebo_GR1 Group (Placebo Comparator): Adults 18 to 50 years of age in Stage 1 (Europe) randomized to receive two doses of altSonflex Placebo, one each at Day 1 and Day 85.
  Interventions: Drug: altSonflex Placebo
- ST1_Adults_Dose C_GR1 Group (Experimental): Adults 18 to 50 years of age in Stage 1 (Europe) randomized to receive two doses of altSonflex1-2-3 Dose C vaccine, one each at Day 1 and Day 85.
  Interventions: Biological: altSonflex1-2-3 Dose C
- ST1_Adults_Placebo_GR2 Group (Placebo Comparator): Adults 18 to 50 years of age in Stage 1 (Europe) randomized to receive two doses of altSonflex Placebo, one each at Day 1 and Day 169.
  Interventions: Drug: altSonflex Placebo
- ST1_Adults_Dose C_GR2 Group (Experimental): Adults 18 to 50 years of age in Stage 1 (Europe) randomized to receive two doses of altSonflex1-2-3 Dose C vaccine, one each at Day 1 and Day 169.
  Interventions: Biological: altSonflex1-2-3 Dose C
- ST2_Adults_Control C Group (Active Comparator): Adults 18 to 50 years of age in Stage 2 (Africa) randomized to receive one dose of GSK's Meningococcal A, C, Y and W-135 conjugate vaccine at Day 1 and one dose of GSK's Tetanus toxoid, reduced diphtheria toxoid and acellular pertussis vaccine at Day 85.
  Interventions: Biological: GSK's Meningococcal A, C, Y and W-135 conjugate vaccine; Combination Product: GSK's Tetanus toxoid, reduced diphtheria toxoid and acellular pertussis vaccine
- ST2_Adults_Dose C Group (Experimental): Adults 18 to 50 years of age in Stage 2 (Africa) randomized to receive two doses of altSonflex1-2-3 Dose C vaccine, one each at Day 1 and Day 85.
  Interventions: Biological: altSonflex1-2-3 Dose C
- ST2_Children_Control B Group (Active Comparator): Children 24 to 59 months of age in Stage 2 (Africa) randomized to receive one dose of GSK's Meningococcal A, C, Y and W-135 conjugate vaccine at Day 1 and one dose of Sanofi Pasteur's Typhoid Vi polysaccharide vaccine at Day 85. This group is a control group for children receiving altSonflex1-2-3 Dose B vaccine.
  Interventions: Biological: GSK's Meningococcal A, C, Y and W-135 conjugate vaccine; Combination Product: Sanofi Pasteur's Typhoid Vi polysaccharide vaccine
- ST2_Children_Dose B Group (Experimental): Children 24 to 59 months of age in Stage 2 (Africa) randomized to receive two doses of altSonflex1-2-3 Dose B vaccine, one each at Day 1 and Day 85.
  Interventions: Biological: altSonflex1-2-3 Dose B
- ST2_Children_Control C Group (Active Comparator): Children 24 to 59 months of age in Stage 2 (Africa) randomized to receive one dose of GSK's Meningococcal A, C, Y and W-135 conjugate vaccine at Day 1 and one dose of Sanofi Pasteur's Typhoid Vi polysaccharide vaccine at Day 85. This group is a control group for children receiving altSonflex1-2-3 Dose C vaccine.
  Interventions: Biological: GSK's Meningococcal A, C, Y and W-135 conjugate vaccine; Combination Product: Sanofi Pasteur's Typhoid Vi polysaccharide vaccine
- ST2_Children_Dose C Group (Experimental): Children 24 to 59 months of age in Stage 2 (Africa) randomized to receive two doses of altSonflex1-2-3 Dose C vaccine, one each at Day 1 and Day 85.
  Interventions: Biological: altSonflex1-2-3 Dose C
- ST2_Infants_Control A_Safety Group (Active Comparator): Infants 9 months of age in Stage 2 (Africa), part of the safety cohort, randomized to receive two doses of GSK's Meningococcal A, C, Y and W-135 conjugate vaccine, one each at Day 1 and Day 85, and one dose of GSK's Diphtheria, tetanus, pertussis, hepatitis B, poliomyelitis (inactivated), and Haemophilus influenzae type b vaccine at Day 253. These infants also receive two doses of Serum Institute of India's Measles and rubella vaccine, one each at Day 29 and Day 281, as concomitant vaccination. This group is a control group for infants receiving altSonflex1-2-3 Dose A vaccine.
  Interventions: Biological: GSK's Meningococcal A, C, Y and W-135 conjugate vaccine; Combination Product: GSK's Diphtheria, tetanus, pertussis, hepatitis B, poliomyelitis (inactivated), and Haemophilus influenzae type b vaccine; Biological: Serum Institute of India's Measles and rubella vaccine
- ST2_Infants_Dose A_Safety Group (Experimental): Infants 9 months of age in Stage 2 (Africa), part of the safety cohort, randomized to receive three doses of altSonflex1-2-3 Dose A, one each at Day 1, Day 85 and Day 253. These infants also receive two doses of Serum Institute of India's Measles and rubella vaccine, one each at Day 29 and Day 281, as concomitant vaccination.
  Interventions: Biological: altSonflex1-2-3 Dose A; Biological: Serum Institute of India's Measles and rubella vaccine
- ST2_Infants_Control B_Safety Group (Active Comparator): Infants 9 months of age in Stage 2 (Africa), part of the safety cohort, randomized to receive two doses of GSK's Meningococcal A, C, Y and W-135 conjugate vaccine, one each at Day 1 and Day 85, and one dose of GSK's Diphtheria, tetanus, pertussis, hepatitis B, poliomyelitis (inactivated), and Haemophilus influenzae type b vaccine at Day 253. These infants also receive two doses of Serum Institute of India's Measles and rubella vaccine, one each at Day 29 and Day 281, as concomitant vaccination. This group is a control group for infants receiving altSonflex1-2-3 Dose B vaccine.
  Interventions: Biological: GSK's Meningococcal A, C, Y and W-135 conjugate vaccine; Combination Product: GSK's Diphtheria, tetanus, pertussis, hepatitis B, poliomyelitis (inactivated), and Haemophilus influenzae type b vaccine; Biological: Serum Institute of India's Measles and rubella vaccine
- ST2_Infants_Dose B_Safety Group (Experimental): Infants 9 months of age in Stage 2 (Africa), part of the safety cohort, randomized to receive three doses of altSonflex1-2-3 Dose B vaccine, one each at Day 1, Day 85 and Day 253. These infants also receive two doses of Serum Institute of India's Measles and rubella vaccine, one each at Day 29 and Day 281, as concomitant vaccination.
  Interventions: Biological: altSonflex1-2-3 Dose B; Biological: Serum Institute of India's Measles and rubella vaccine
- ST2_Infants_Control C_Safety Group (Active Comparator): Infants 9 months of age in Stage 2 (Africa), part of the safety cohort, randomized to receive two doses of GSK's Meningococcal A, C, Y and W-135 conjugate vaccine, one each at Day 1 and Day 85, and one dose of GSK's Diphtheria, tetanus, pertussis, hepatitis B, poliomyelitis (inactivated), and Haemophilus influenzae type b vaccine at Day 253. These infants also receive two doses of Serum Institute of India's Measles and rubella vaccine, one each at Day 29 and Day 281, as concomitant vaccination. This group is a control group for infants receiving altSonflex1-2-3 Dose C vaccine.
  Interventions: Biological: GSK's Meningococcal A, C, Y and W-135 conjugate vaccine; Combination Product: GSK's Diphtheria, tetanus, pertussis, hepatitis B, poliomyelitis (inactivated), and Haemophilus influenzae type b vaccine; Biological: Serum Institute of India's Measles and rubella vaccine
- ST2_Infants_Dose C_Safety Group (Experimental): Infants 9 months of age in Stage 2 (Africa), part of the safety cohort, randomized to receive three doses of altSonflex1-2-3 Dose C vaccine, one each at Day 1, Day 85 and Day 253. These infants also receive two doses of Serum Institute of India's Measles and rubella vaccine, one each at Day 29 and Day 281, as concomitant vaccination.
  Interventions: Biological: altSonflex1-2-3 Dose C; Biological: Serum Institute of India's Measles and rubella vaccine
- ST2_Infants_Control_Dose find Group (Active Comparator): Infants 9 months of age in Stage 2 (Africa), part of the dose-finding cohort, randomized to receive two doses of GSK's Meningococcal A, C, Y and W-135 conjugate vaccine, one each at Day 1 and Day 85, and one dose of GSK's Diphtheria, tetanus, pertussis, hepatitis B, poliomyelitis (inactivated), and Haemophilus influenzae type b vaccine at Day 253.
  These infants also receive two doses of Serum Institute of India's Measles and rubella vaccine, one each at Day 1 and Day 253, as concomitant vaccination. This group is a control group for infants in dose-finding groups receiving either altSonflex1-2-3 Dose A, Dose B or Dose C vaccine.
  Interventions: Biological: GSK's Meningococcal A, C, Y and W-135 conjugate vaccine; Combination Product: GSK's Diphtheria, tetanus, pertussis, hepatitis B, poliomyelitis (inactivated), and Haemophilus influenzae type b vaccine; Biological: Serum Institute of India's Measles and rubella vaccine
- ST2_Infants_Dose A_Dose find Group (Experimental): Infants 9 months of age in Stage 2 (Africa), part of the dose-finding cohort, randomized to receive three doses of altSonflex1-2-3 Dose A vaccine, one each at Day 1, Day 85 and Day 253. These infants also receive two doses of Serum Institute of India's Measles and rubella vaccine, one each at Day 1 and Day 253, as concomitant vaccination.
  Interventions: Biological: altSonflex1-2-3 Dose A; Biological: Serum Institute of India's Measles and rubella vaccine
- ST2_Infants_Dose B_Dose find Group (Experimental): Infants 9 months of age in Stage 2 (Africa), part of the dose-finding cohort, randomized to receive three doses of altSonflex1-2-3 Dose B vaccine, one each at Day 1, Day 85 and Day 253. These infants also receive two doses of Serum Institute of India's Measles and rubella vaccine, one each at Day 1 and Day 253, as concomitant vaccination.
  Interventions: Biological: altSonflex1-2-3 Dose B; Biological: Serum Institute of India's Measles and rubella vaccine
- ST2_Infants_Dose C_Dose find Group (Experimental): Infants 9 months of age in Stage 2 (Africa), part of the dose-finding cohort, randomized to receive three doses of altSonflex1-2-3 Dose C vaccine, one each at Day 1, Day 85 and Day 253. These infants also receive two doses of Serum Institute of India's Measles and rubella vaccine, one each at Day 1 and Day 253, as concomitant vaccination.
  Interventions: Biological: altSonflex1-2-3 Dose C; Biological: Serum Institute of India's Measles and rubella vaccine

INTERVENTIONS:
Drug: altSonflex Placebo — 2 doses of altSonflex Placebo, administered intramuscularly, in the non-dominant arm, either at Day 1 and Day 85 or at Day 1 and Day 169 (depending on the vaccination schedule) to adults in the ST1_Adults_Placebo_GR1 and ST1_Adults_Placebo_GR2 groups in Stage 1 (Europe).
  Arms: ST1_Adults_Placebo_GR1 Group; ST1_Adults_Placebo_GR2 Group
Biological: altSonflex1-2-3 Dose C — 2 doses of altSonflex1-2-3 Dose C administered intramuscularly, in the non-dominant arm, at Day 1 and Day 85 to adults in the ST1_Adults_Dose C_GR1 and ST2_Adults_Dose C groups in Stage 1 and 2 (Europe and Africa) and children in the ST2_Children_Dose C group in Stage 2 (Africa), and at Day 1 and Day 169 to adults in the ST1_Adults_Dose C_GR2 group in Stage 1 (Europe); 3 doses of altSonflex1-2-3 Dose C administered intramuscularly, in the non-dominant arm, at Day 1, Day 85 and Day 253 to infants in the ST2_Infants_Dose C_Safety and ST2_Infants_Dose C_Dose find groups in Stage 2 (Africa).
  Other Names: Shigella vaccine
  Arms: ST1_Adults_Dose C_GR1 Group; ST1_Adults_Dose C_GR2 Group; ST2_Adults_Dose C Group; ST2_Children_Dose C Group; ST2_Infants_Dose C_Dose find Group; ST2_Infants_Dose C_Safety Group
Biological: altSonflex1-2-3 Dose B — 2 doses of altSonflex1-2-3 Dose B administered intramuscularly, in the non-dominant arm, at Day 1 and Day 85 to children in the ST2_Children_Dose B group in Stage 2 (Africa); 3 doses of altSonflex1-2-3 Dose B administered intramuscularly, in the non-dominant arm, at Day 1, Day 85 and Day 253 to infants in the ST2_Infants_Dose B_Safety and ST2_Infants_Dose B_Dose find groups in Stage 2 (Africa).
  Other Names: Shigella vaccine
  Arms: ST2_Children_Dose B Group; ST2_Infants_Dose B_Dose find Group; ST2_Infants_Dose B_Safety Group
Biological: altSonflex1-2-3 Dose A — 3 doses of altSonflex1-2-3 Dose A administered intramuscularly, in the non-dominant arm, at Day 1, Day 85 and Day 253 to infants in the ST2_Infants_Dose A_Safety and ST2_Infants_Dose A_Dose find groups in Stage 2 (Africa).
  Other Names: Shigella vaccine
  Arms: ST2_Infants_Dose A_Dose find Group; ST2_Infants_Dose A_Safety Group
Biological: GSK's Meningococcal A, C, Y and W-135 conjugate vaccine — 1 dose of GSK's Meningococcal A, C, Y and W-135 conjugate vaccine administered intramuscularly, in the non-dominant arm, at Day 1 to adults in the ST2_Adults_Control C group and children in the ST2_Children_Control B and ST2_Children_Control C groups in Stage 2 (Africa); 2 doses of GSK's Meningococcal A, C, Y and W-135 conjugate vaccine administered intramuscularly, in the non-dominant arm, at Day 1 and Day 85 to infants in the ST2_Infants_Control A_Safety, ST2_Infants_Control B_Safety, ST2_Infants_Control C_Safety and ST2_Infants_Control_Dose find groups in Stage 2 (Africa).
  Other Names: MENVEO
  Arms: ST2_Adults_Control C Group; ST2_Children_Control B Group; ST2_Children_Control C Group; ST2_Infants_Control A_Safety Group; ST2_Infants_Control B_Safety Group; ST2_Infants_Control C_Safety Group; ST2_Infants_Control_Dose find Group
Combination Product: GSK's Tetanus toxoid, reduced diphtheria toxoid and acellular pertussis vaccine — 1 dose of GSK's Tetanus toxoid, reduced diphtheria toxoid and acellular pertussis vaccine administered intramuscularly, in the non-dominant arm, at Day 85 to adults in the ST2_Adults_Control C group in Stage 2 (Africa).
  Other Names: BOOSTRIX
  Arms: ST2_Adults_Control C Group
Combination Product: GSK's Diphtheria, tetanus, pertussis, hepatitis B, poliomyelitis (inactivated), and Haemophilus influenzae type b vaccine — 1 dose of GSK's Diphtheria, tetanus, pertussis, hepatitis B, poliomyelitis (inactivated), and Haemophilus influenzae type b vaccine administered intramuscularly, in the non-dominant arm, at Day 253 to infants in the ST2_Infants_Control A_Safety, ST2_Infants_Control B_Safety, ST2_Infants_Control C_Safety and ST2_Infants_Control_Dose find groups in Stage 2 (Africa).
  Other Names: INFANRIX Hexa
  Arms: ST2_Infants_Control A_Safety Group; ST2_Infants_Control B_Safety Group; ST2_Infants_Control C_Safety Group; ST2_Infants_Control_Dose find Group
Combination Product: Sanofi Pasteur's Typhoid Vi polysaccharide vaccine — 1 dose of Sanofi Pasteur's Typhoid Vi polysaccharide vaccine administered intramuscularly, in the non-dominant arm, at Day 85 to children in the ST2_Children_Control B and ST2_Children_Control C groups in Stage 2 (Africa).
  Other Names: TYPHIM VI
  Arms: ST2_Children_Control B Group; ST2_Children_Control C Group
Biological: Serum Institute of India's Measles and rubella vaccine — 2 doses of Serum Institute of India's Measles and rubella vaccine administered subcutaneously, in the non-dominant arm, at Day 29 and Day 281 to infants in the safety groups, and at Day 1 and Day 253 to infants in the dose-finding groups, in Stage 2 (Africa).
  Other Names: MR-VAC
  Arms: ST2_Infants_Control A_Safety Group; ST2_Infants_Control B_Safety Group; ST2_Infants_Control C_Safety Group; ST2_Infants_Control_Dose find Group; ST2_Infants_Dose A_Dose find Group; ST2_Infants_Dose A_Safety Group; ST2_Infants_Dose B_Dose find Group; ST2_Infants_Dose B_Safety Group; ST2_Infants_Dose C_Dose find Group; ST2_Infants_Dose C_Safety Group

SUMMARY:
The aim of the current clinical study is to evaluate, for the first time in humans (FTIH), the safety and immunogenicity of the altSonflex1-2-3 candidate vaccine against S. sonnei and S. flexneri serotypes 1b, 2a, and 3a. The vaccine will be first administered in adults 18 to 50 years of age in Europe. Subsequently, the vaccine will be administered to a shigellosis-endemic population in Africa, first in adults 18 to 50 years of age, then in children 24 to 59 months of age, finally in infants 9 months of age. Infants will also receive a third vaccination. Three different doses of the vaccine [low (Dose A), medium (Dose B), and high (Dose C) amounts of antigen] will be evaluated using an age de-escalation approach (from least vulnerable adult population to most vulnerable paediatric population). The results of this study will allow the selection of the most appropriate dose for further vaccine development in infants 9 months of age, which is the main target age group for this vaccine.

ELIGIBILITY:
Inclusion Criteria:

All participants:

* Participants and/or participants' parent(s)/legally acceptable representative(s) LAR(s), who, in the opinion of the investigator, can and will comply with the requirements of the protocol (e.g. completion of the diary cards, return for follow-up visits).
* Written or witnessed/thumb printed informed consent obtained from the participant/parent(s)/LAR(s) of the participant prior to performance of any study specific procedure.
* Healthy participants as established by medical history, clinical examination, and laboratory assessment.
* Participants satisfying all screening requirements.
* Participants seronegative for hepatitis B, and hepatitis C.
* Participants negative for human leukocyte antigen B27 (HLA-B27).

Adults 18 to 50 years of age:

* A male or female between, and including, 18 and 50 years of age at the time of the first study intervention administration.
* Female participants of non-childbearing potential may be enrolled in the study. Non-childbearing potential is defined as pre-menarche, current bilateral tubal ligation or occlusion, hysterectomy, bilateral ovariectomy or post-menopause.
* Female participants of childbearing potential may be enrolled in the study, if the participant:

  - has practiced adequate contraception for 1 month prior to study intervention administration, and

  - has a negative pregnancy test on the day of study intervention administration, and
  * has agreed to continue adequate contraception during the entire treatment period and for 1 month after completion of the study intervention administration series.
* Participants seronegative for human immunodeficiency virus (HIV).

Children 24 to 59 months of age:

* A male or female between, and including, 24 and 59 months of age at the time of first vaccination.
* Normal nutritional Z score (-2 standard deviation or greater).
* Previously completed routine childhood vaccinations to the best knowledge of the participant's parent(s)/LAR(s).
* Born after gestation period of ≥37 weeks.
* Participants seronegative for HIV.

Infants 9 months of age:

* A male or female 9 months of age at the time of first vaccination.
* Normal nutritional Z score (-2 standard deviations or greater).
* Previously completed routine childhood vaccinations to the best knowledge of the participant's parent(s)/LAR(s).
* Born after a gestation period of ≥37 weeks.
* Participants negative for HIV as confirmed by deoxyribonucleic acid (DNA) polymerase chain reaction (PCR) testing.

Exclusion Criteria:

All participants:

* Known exposure to Shigella during lifetime of the participant as confirmed during interview with the participant or documented by patient records (e.g., history of microbiologically-confirmed Shigella infection), recent travel* (within 2 years) to a country where Shigella or other enteric infections are endemic, or recent occupation* (within 3 years) involving Shigella species.

  *Exclusion due to travel or occupation is applicable only to Adults 18 to 50 years of age in Europe (Stage 1).
* Progressive, unstable or uncontrolled clinical conditions.
* History (known or suspected) of any reaction or hypersensitivity likely to be exacerbated by any component of the study vaccine.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination (no laboratory testing required).
* Hypersensitivity, including allergy, to medicinal products or medical equipment whose use is foreseen in this study.
* Clinical conditions representing a contraindication to IM vaccination and blood draws.
* Any behavioural or cognitive impairment or psychiatric disease that, in the opinion of the investigator, may interfere with the participant's ability to participate in the study.
* Acute disease and/or fever (defined as temperature ≥38.0°C) at the time of enrolment*.

  * The participant can still be enrolled into the study at a time when the acute disease and/or fever has resolved.
* Any clinically significant haematological and/or biochemical laboratory abnormality.
* Confirmed positive COVID-19 test during the period starting 30 days before the first administration of study vaccines (Day -30 to Day 1).
* Any other clinical condition that, in the opinion of the investigator, might pose additional risk to the participant due to participation in the study.
* Administration of long-acting immune-modifying drugs at any time during the study period (e.g. infliximab).
* Prior receipt of an experimental Shigella vaccine or live Shigella challenge.
* Use of any investigational or non-registered product (drug, vaccine or medical device)* other than the study vaccine during the period starting 30 days before the first dose of study intervention (Day -30 to Day 1), or planned use during the study period.

  *Use of herbs and traditional treatments is not considered an exclusion criterion
* A vaccine not foreseen* by the Study Protocol administered during the period starting at -21 days before the first dose (-28 days in the case of live vaccines) and ending after the last dose of study intervention administration**.

  *Vaccines allowed by the Protocol include flu and COVID-19 vaccines in all participants and EPI vaccines in children and infants.

  **In case of emergency mass vaccination, the time period above can be reduced.
* Concurrently participating in another clinical study, at any time during the study period, in which the participant has been or will be exposed to an investigational or a non-investigational intervention (drug or invasive medical device).
* Any study personnel or immediate dependents, family, or household member.

Adults 18 to 50 years of age:

* Acute or chronic illness, clinically significant pulmonary, cardiovascular, hepatic or renal functional abnormality, as determined by physical examination or laboratory screening tests.
* Chronic administration (defined as more than 14 days in total) of immunosuppressants or other immune-modifying drugs during the period starting 3 months prior to the first vaccine study intervention. For corticosteroids, this will mean prednisone equivalent ≥20 mg/day for adult participants. Inhaled and topical steroids are allowed.
* Pregnant or lactating female.
* Female planning to become pregnant or planning to discontinue contraceptive precautions.
* History of or current chronic alcohol consumption and/or drug abuse.

Adults 18 to 50 years of age and Children 24 to 59 months age:

• Administration of immunoglobulins and/or any blood products or plasma derivatives, or bone marrow transplantation, during the period starting 3 months before the first dose of study vaccine or planned administration during the study period.

Children 24 to 59 months of age and infants 9 months of age:

* Acute or chronic clinically significant pulmonary, cardiovascular, hepatic or renal functional abnormality, as determined by physical examination or laboratory screening tests.
* Chronic administration (defined as more than 14 days in total) of immunosuppressants or other immune-modifying drugs during the period starting 3 months prior to the first vaccine dose. For corticosteroids, this will mean prednisone ≥0.5 mg/kg/day or 20 mg/day whichever is the maximum dose for paediatric participants. Inhaled and topical steroids are allowed.
* Child in care.

Infants 9 months of age:

• Administration of immunoglobulins and/or any blood products or plasma derivatives, or bone marrow transplantation, from birth or planned administration during the study period.

Ages: 9 Months to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 551 (Actual)
Dates: Start 2021-10-06 (Actual); Primary Completion 2025-06-24 (Actual); Study Completion 2025-06-24 (Actual)

PRIMARY OUTCOMES:
Anti-serotype specific Shigella lipopolysaccharide (LPS)/O-Antigen (OAg) serum immunoglobulin G (IgG) geometric mean concentrations (GMCs) in infants 9 months of age in Africa | At Day 281 (28 days after the third study intervention administration)
  Anti-serotype specific Shigella LPS/OAg serum IgG GMCs are measured by GSK Vaccines Institute for Global Health (GVGH) enzyme-linked immunosorbent assay (ELISA) and expressed in ELISA units per milliliter (EU/mL) of serum.
Number of adults 18 to 50 years of age in Europe with solicited administration site events | During 7 days after each study intervention administration (study interventions administered at Day 1 and Day 85/Day 169)
  The solicited administration site events are pain, redness, and swelling.
Number of adults 18 to 50 years of age in Europe with solicited systemic events | During 7 days after each study intervention administration (study interventions administered at Day 1 and Day 85/Day 169)
  The solicited systemic event is fever. Fever is defined as temperature equal to or above (≥) 38.0°C. The preferred location for measuring temperature is the axilla for all participants.
Number of adults 18 to 50 years of age in Europe with unsolicited adverse events (AEs) | During 28 days after each study intervention administration (study interventions administered at Day 1 and Day 85/Day 169)
  An unsolicited AE is an AE reported in addition to those solicited during the clinical study. Also, any 'solicited' symptom with onset outside the specified period of follow-up for solicited symptoms is reported as an unsolicited adverse event.
Number of adults 18 to 50 years of age in Europe with serious adverse events (SAEs) | During the entire study participation period [Day 1 to Day 113 (for ST1_Adults_Placebo_GR1 and ST1_Adults_Dose C_GR1 groups)/Day 197 (for ST1_Adults_Placebo_GR2 and ST1_Adults_Dose C_GR2 groups)
  An SAE is defined as any untoward medical occurrence that results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect in the offspring of a study participant, results in abnormal pregnancy outcomes or any other situation based on appropriate medical or scientific judgement.
Number of adults 18 to 50 years of age in Europe with deviations from normal values of haematological, renal, and hepatic panel test results at Day 8 (7 days after the first study intervention administration) | At Day 8 (7 days after the first study intervention administration)
  Panel tests include measures of leukocytes, erythrocytes, haemoglobin, haematocrit, platelets, eosinophils, basophils, neutrophils, monocytes, lymphocytes, creatinine, blood urea, sodium, potassium, aspartate aminotransferase (AST) and alanine aminotransferase (ALT).
Number of adults 18 to 50 years of age in Europe with deviations from normal values of haematological, renal, and hepatic panel test results at Day 92/Day 176 (7 days after the second study intervention administration) | At Day 92 (for ST1_Adults_Placebo_GR1 and ST1_Adults_Dose C_GR1 groups)/Day 176 (for ST1_Adults_Placebo_GR2 and ST1_Adults_Dose C_GR2 groups) (7 days after the second study intervention administration)
  Panel tests include measures of leukocytes, erythrocytes, haemoglobin, haematocrit, platelets, eosinophils, basophils, neutrophils, monocytes, lymphocytes, creatinine, blood urea, sodium, potassium, aspartate aminotransferase (AST) and alanine aminotransferase (ALT).
Number of adults 18 to 50 years of age in Africa with solicited administration site events | During 7 days after each study intervention administration (study interventions administered at Day 1 and Day 85)
  The solicited administration site events are pain, redness, and swelling.
Number of adults 18 to 50 years of age in Africa with solicited systemic events | During 7 days after each study intervention administration (study interventions administered at Day 1 and Day 85)
  The solicited systemic event is fever. Fever is defined as temperature ≥ 38.0°C. The preferred location for measuring temperature is the axilla for all participants.
Number of adults 18 to 50 years of age in Africa with unsolicited AEs | During 28 days after each study intervention administration (study interventions administered at Day 1 and Day 85)
  An unsolicited AE is an AE reported in addition to those solicited during the clinical study. Also, any 'solicited' symptom with onset outside the specified period of follow-up for solicited symptoms is reported as an unsolicited adverse event.
Number of adults 18 to 50 years of age in Africa with SAEs | During the entire study participation (Day 1 to Day 113)
  An SAE is defined as any untoward medical occurrence that results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect in the offspring of a study participant, results in abnormal pregnancy outcomes or any other situation based on appropriate medical or scientific judgement.
Number of adults 18 to 50 years of age in Africa with deviations from normal values of haematological, renal, and hepatic panel test results at Day 8 (7 days after the first study intervention administration) | At Day 8 (7 days after the first study intervention administration)
  Panel tests include measures of leukocytes, erythrocytes, haemoglobin, haematocrit, platelets, eosinophils, basophils, neutrophils, monocytes, lymphocytes, creatinine, blood urea, sodium, potassium, AST, and ALT.
Number of adults 18 to 50 years of age in Africa with deviations from normal values of haematological, renal, and hepatic panel test results at Day 92 (7 days after the second study intervention administration) | At Day 92 (7 days after the second study intervention administration)
  Panel tests include measures of leukocytes, erythrocytes, haemoglobin, haematocrit, platelets, eosinophils, basophils, neutrophils, monocytes, lymphocytes, creatinine, blood urea, sodium, potassium, AST, and ALT.
Number of children 24 to 59 months of age in Africa with solicited administration site events | During 7 days after each study intervention administration (study interventions administered at Day 1 and Day 85)
  The solicited administration site events are pain, redness, and swelling.
Number of children 24 to 59 months of age in Africa with solicited systemic events | During 7 days after each study intervention administration (study interventions administered at Day 1 and Day 85)
  The solicited systemic event is fever. Fever is defined as temperature ≥ 38.0°C. The preferred location for measuring temperature is the axilla for all participants.
Number of children 24 to 59 months of age in Africa with unsolicited AEs | During 28 days after each study intervention administration (study interventions administered on Day 1 and Day 85)
  An unsolicited AE is an AE reported in addition to those solicited during the clinical study. Also, any 'solicited' symptom with onset outside the specified period of follow-up for solicited symptoms is reported as an unsolicited adverse event.
Number of children 24 to 59 months of age in Africa with SAEs | During the entire study participation period (Day 1 to Day 113)
  An SAE is defined as any untoward medical occurrence that results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in disability/incapacity or any other situation based on appropriate medical or scientific judgement.
Number of children 24 to 59 months of age in Africa with deviations from normal values of haematological, renal, and hepatic panel test results at Day 8 (7 days after the first study intervention administration) | At Day 8 (7 days after the first study intervention administration)
  Panel tests include measures of leukocytes, erythrocytes, haemoglobin, haematocrit, platelets, eosinophils, basophils, neutrophils, monocytes, lymphocytes, creatinine, blood urea, sodium, potassium, AST, and ALT.
Number of children 24 to 59 months of age in Africa with deviations from normal values of haematological, renal, and hepatic panel test results at Day 92 (7 days after the second study intervention administration) | At Day 92 (7 days after the second study intervention administration)
  Panel tests include measures of leukocytes, erythrocytes, haemoglobin, haematocrit, platelets, eosinophils, basophils, neutrophils, monocytes, lymphocytes, creatinine, blood urea, sodium, potassium, AST, and ALT.
Number of infants 9 months of age in Africa with solicited administration site events | During 7 days after each study intervention administration (study interventions administered at Day 1, Day 85 and Day 253)
  The solicited administration site events are pain, redness and swelling.
Number of infants 9 months of age in Africa with solicited systemic events | During 7 days after each study intervention administration (study interventions administered at Day 1, Day 85 and Day 253)
  The solicited systemic event is fever. Fever is defined as temperature ≥ 38.0°C. The preferred location for measuring temperature is the axilla for all participants.
Number of infants 9 months of age in Africa with unsolicited AEs | During 28 days after each study intervention administration (study intervention administered at Day 1, Day 85 and Day 253)
  An unsolicited AE is an AE reported in addition to those solicited during the clinical study. Also, any 'solicited' symptom with onset outside the specified period of follow-up for solicited symptoms is reported as an unsolicited adverse event.
Number of infants 9 months of age in Africa with SAEs | During the entire study participation period (Day 1 to Day 281)
  An SAE is defined as any untoward medical occurrence that results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in disability/incapacity or any other situation based on appropriate medical or scientific judgement.
Number of infants 9 months of age in Africa with deviations from normal values of haematological, renal, and hepatic panel test results at Day 8 (7 days after the first study intervention administration) | At Day 8 (7 days after the first study intervention administration)
  Panel tests include measures of leukocytes, erythrocytes, haemoglobin, haematocrit, platelets, eosinophils, basophils, neutrophils, monocytes, lymphocytes, creatinine, blood urea, sodium, potassium, AST, and ALT.
Number of infants 9 months of age in Africa with deviations from normal values of haematological, renal, and hepatic panel test results at Day 92 (7 days after the second study intervention administration) | At Day 92 (7 days after the second study intervention administration)
  Panel tests include measures of leukocytes, erythrocytes, haemoglobin, haematocrit, platelets, eosinophils, basophils, neutrophils, monocytes, lymphocytes, creatinine, blood urea, sodium, potassium, AST, and ALT.
Number of infants 9 months of age in Africa with deviations from normal values of haematological, renal, and hepatic panel test results at Day 260 (7 days after the third study intervention administration) | At Day 260 (7 days after the third study intervention administration)
  Panel tests include measures of leukocytes, erythrocytes, haemoglobin, haematocrit, platelets, eosinophils, basophils, neutrophils, monocytes, lymphocytes, creatinine, blood urea, sodium, potassium, AST, and ALT.

SECONDARY OUTCOMES:
Anti-serotype specific Shigella LPS/OAg serum IgG GMCs in adults 18 to 50 years of age in Europe | At Day 1 and Day 85/Day 169 (before each study intervention administration), at Day 15 (14 days after the first study intervention administration) and at Day 29 and Day 113/Day197 (28 days after each study intervention administration)
  Anti-serotype specific Shigella LPS/OAg serum IgG GMCs are measured by GVGH ELISA and expressed in EU/mL of serum.
Anti-serotype specific Shigella LPS/OAg serum IgG GMCs in adults 18 to 50 years of age in Africa | At Day 1 and Day 85 (before each study intervention administration) and at Day 29 and Day 113 (28 days after each study intervention administration)
  Anti-serotype specific Shigella LPS/OAg serum IgG GMCs are measured by GVGH ELISA and expressed in EU/mL of serum.
Anti-serotype specific Shigella LPS/OAg serum IgG GMCs in children 24 to 59 months of age in Africa | At Day 1 and Day 85 (before each study intervention administration) and at Day 29 and Day 113 (28 days after each study intervention administration)
  Anti-serotype specific Shigella LPS/OAg serum IgG GMCs are measured by GVGH ELISA and expressed in EU/mL of serum.
Anti-serotype specific Shigella LPS/OAg serum IgG GMCs in infants 9 months of age in Africa | At Day 1, Day 85 and Day 253 (before each study intervention administration) and at Day 29, Day 113 and Day 281 (28 days after each study intervention administration)
  Anti-serotype specific Shigella LPS/OAg serum IgG GMCs are measured by GVGH ELISA and expressed in EU/mL of serum.
Number of adults 18 to 50 years of age in Europe achieving a GVGH ELISA level equivalent to ≥1:800 titer against S. sonnei LPS/OAg | At Day 1 and Day 85/Day 169 (before each study intervention administration), at Day 15 (14 days after the first study intervention administration) and at Day 29 and Day 113/Day 197 (28 days after each study intervention administration)
Number of adults 18 to 50 years of age in Africa achieving a GVGH ELISA level equivalent to ≥1:800 titer against S. sonnei LPS/OAg | At Day 1 and Day 85 (before each study intervention administration) and at Day 29 and Day 113 (28 days after each study intervention administration)
Number of children 24 to 59 months of age in Africa achieving a GVGH ELISA level equivalent to ≥1:800 titer against S. sonnei LPS/OAg | At Day 1 and Day 85 (before each study intervention administration) and at Day 29 and Day 113 (28 days after each study intervention administration)
Number of infants 9 months of age in Africa achieving a GVGH ELISA level equivalent to ≥1:800 titer against S. sonnei LPS/OAg | At Day 1, Day 85 and Day 253 (before each study intervention administration) and at Day 29, Day 113 and Day 281 (28 days after each study intervention administration)
Number of adults 18 to 50 years of age in Europe achieving a GVGH ELISA level equivalent to ≥1:1600 titer against S. sonnei LPS/OAg | At Day 1 and Day 85/Day 169 (before each study intervention administration), at Day 15 (14 days after the first study intervention administration) and at Day 29 and Day 113/Day 197 (28 days after each study intervention administration)
Number of adults 18 to 50 years of age in Africa achieving a GVGH ELISA level equivalent to ≥1:1600 titer against S. sonnei LPS/OAg | At Day 1 and Day 85 (before each study intervention administration) and at Day 29 and Day 113 (28 days after each study intervention administration)
Number of children 24 to 59 months of age in Africa achieving a GVGH ELISA level equivalent to ≥1:1600 titer against S. sonnei LPS/OAg | At Day 1 and Day 85 (before each study intervention administration) and at Day 29 and Day 113 (28 days after each study intervention administration)
Number of infants 9 months of age in Africa achieving a GVGH ELISA level equivalent to ≥1:1600 titer against S. sonnei LPS/OAg | At Day 1, Day 85 and Day 253 (before each study intervention administration) and at Day 29, Day 113 and Day 281 (28 days after each study intervention administration)
Number of adults 18 to 50 years of age in Europe showing at least a 4-fold increase in anti-serotype specific Shigella LPS/OAg serum IgG concentrations, as measured by GVGH ELISA | At Day 15 (14 days after first study intervention administration) and at Day 29 and Day 113/197 (28 days after each study intervention administration) compared to Day 1 and Day 85/Day 169 (baseline)
Number of adults 18 to 50 years of age in Africa showing at least a 4-fold increase in anti-serotype specific Shigella LPS/OAg serum IgG concentrations, as measured by GVGH ELISA | At Day 29 and Day 113 (28 days after each study intervention administration) compared to Day 1 and Day 85 (baseline)
Number of children 24 to 59 months of age in Africa showing at least a 4-fold increase in anti-serotype specific Shigella LPS/OAg serum IgG concentrations, as measured by GVGH ELISA | At Day 29 and Day 113 (28 days after each study intervention administration) compared to Day 1 and Day 85 (baseline)
Number of infants 9 months of age in Africa showing at least a 4-fold increase in anti-serotype specific Shigella LPS/OAg serum IgG concentrations, as measured by GVGH ELISA | At Day 29, Day 113 and Day 281 (28 days after each study intervention administration) compared to Day 1, Day 85 and Day 253 (baseline)
Anti-measles IgG concentrations in infants 9 months of age in the dose-finding groups in Africa | At Day 1 (before the first MR-VAC dose administration) and Day 281 (28 days after the second MR-VAC dose administration)
Anti-rubella IgG concentrations in infants 9 months of age in the dose-finding groups in Africa | At Day 1 (before the first MR-VAC dose administration) and Day 281 (28 days after the second MR-VAC dose administration)
Number of infants 9 months of age in the dose-finding groups in Africa achieving anti-measles IgG concentrations of ≥150 mIU/mL and ≥200 mIU/mL | At Day 281 (28 days after the second MR-VAC dose administration)
Number of infants 9 months of age in the dose-finding groups in Africa achieving anti-rubella IgG concentrations of ≥4 IU/mL and ≥10 IU/mL | At Day 281 (28 days after the second MR-VAC dose administration)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- GSK Investigational Site, Ghent, Belgium
- GSK Investigational Site, Kericho, Kenya

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.

REFERENCES:
- [Derived] Leroux-Roels I, Maes C, Mancini F, Jacobs B, Sarakinou E, Alhatemi A, Joye J, Grappi S, Cilio GL, Serry-Bangura A, Vitali CG, Ferruzzi P, Marchetti E, Necchi F, Rappuoli R, De Ryck I, Auerbach J, Colucci AM, Rossi O, Conti V, Scorza FB, Arora AK, Micoli F, Podda A, Nakakana UN; Shigella Project Team. Safety and Immunogenicity of a 4-Component Generalized Modules for Membrane Antigens Shigella Vaccine in Healthy European Adults: Randomized, Phase 1/2 Study. J Infect Dis. 2024 Oct 16;230(4):e971-e984. doi: 10.1093/infdis/jiae273. PMID 38853614